CLINICAL TRIAL: NCT01541085
Title: Ex Vivo Study of Immune-Reconstitution Kinetics in HIV-infected ARV-naive Subjects, With Advanced Disease, Starting a Darunavir/Ritonavir or Efavirenz Based HAART (IMMUNO Study)
Brief Title: An Immunologic Study of Treatment-Naive HIV Patients Starting a Darunavir/Ritonavir- or Efavirenz-Based HAART
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR017920; TMC114HIV0010 (Other: Janssen-Cilag S.p.A., Italy)
Record Dates: First submitted 2011-08-23; First posted 2012-02-29 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Human Immunodeficiency Virus; HIV
Keywords: Human Immunodeficiency Virus; HIV; Highly Active Antiretroviral Therapy; HAART; Darunavir; Ritonavir; Efavirenz; Kinetics; Immunological Recovery
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Darunavir; Ritonavir; efavirenz

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Darunavir/Ritonavir (DRV/r)
  Interventions: Drug: Darunavir/Ritonavir (DRV/r)
- Efavirenz (EFV)
  Interventions: Drug: Efavirenz (EFV)

INTERVENTIONS:
Drug: Darunavir/Ritonavir (DRV/r) — Darunavir/Ritonavir (DRV/r) + Tenofovir/Emtricitabina regimen
  Groups: Darunavir/Ritonavir (DRV/r)
Drug: Efavirenz (EFV) — Efavirenz (EFV) + Tenofovir/Emtricitabina regimen
  Groups: Efavirenz (EFV)

SUMMARY:
The purpose of this study is to study the kinetics (study of the rate of change) of immune recovery quality and function in stored plasma blood samples of treatment-naive (not previously treated with antiretroviral drugs) patients with advanced human immunodeficiency virus (HIV) infection starting a Darunavir/Ritonavir- or Efavirenz-based highly active antiretroviral therapy (HAART) regimen.

DETAILED DESCRIPTION:
This is an ex-vivo study (study which takes place outside the organism and records immune parameters from stored blood and cells of a defined population without any intervention by the researcher) to evaluate the kinetics (study of the rate of change) of immune recovery quality and function in stored plasma blood samples of treatment-naive (not previously treated with antiretroviral drugs) patients with advanced human immunodeficiency virus (HIV) infection starting a Darunavir/Ritonavir (DRV/r)- or Efavirenz (EFV)-based highly active antiretroviral therapy (HAART) regimen. In previously stored plasma blood samples, the role of DRV/r compared with EFV in reducing T-lymphocyte activation, DRV/r compared with EFV in recovering T-lymphocyte immune phenotype in peripheral blood and thymic production, and DRV/r compared with EFV in recovering T-lymphocyte function (functional immunity) will be studied. Blood samples will be analyzed before (baseline) and up to 48 weeks after initiating HAART.

Each patient will receive orally administered (given by mouth) regimens of either Darunavir/Ritonavir (DRV/r) + Tenofovir/Emtricitabina or Efavirenz (EFV) + Tenofovir/Emtricitabina.

ELIGIBILITY:
Inclusion Criteria:

* Documented human immunodeficiency (HIV)-1 infection
* At baseline plasma blood sampling, has never received antiretroviral therapy
* Attending the Clinic of Infectious Diseases of the University of Milan at San Paolo Hospital
* Asymptomatic (demonstrating no acquired immunodeficiency syndrome [AIDS]-defining symptoms) at Baseline, Week 12, and Week 24
* CD4 cell count >50 to <250/mm3 at Baseline
* Receiving treatment with either Darunavir/Ritonavir + Tenofovir/Emtricitabina or Efavirenz + Tenofovir/Emtricitabina highly active antiretroviral therapy (HAART) regimens at Week 12, Week 24, and Week 48 plasma blood sampling.

Exclusion Criteria is not defined in protocol.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Antiretroviral treatment-naive patients with advanced HIV infection starting a Darunavir/Ritonavir - or Efavirenz-based HAART regimen. Patients with advanced HIV infection are defined by a treatment-naïve CD4+ cell count >50 to <250 cells/mm3.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2011-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change (>=10%) in the proportion of activated HLA-DR+CD38+CD8+ T-cells | Baseline and Week 24

SECONDARY OUTCOMES:
Change (>=10%) in the proportion of activated HLA-DR+CD38+CD8+ T-cells | Baseline, Week 12, and Week 48
Change in peripheral T-lymphocyte immune phenotype | Baseline, Week 12, Week 24 and Week 48
Change in peripheral T-lymphocyte turnover | Baseline, Week 12, Week 24 and Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag S.p.A., Italy Clinical Trial, Study Director — Janssen-Cilag S.p.A.